CLINICAL TRIAL: NCT03903718
Title: A Phase 1/2a Clinical Study to Evaluate the Efficacy of MEDI8852 in the Treatment of Influenza in Adults Challenged With a Wild-Type Influenza Strain
Brief Title: Evaluation of the Safety and Efficacy of a Monoclonal Antibody to Treat Influenza
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to delay in site enrollment timelines
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6000C00004
Record Dates: First submitted 2019-03-22; First posted 2019-04-04 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Influenza
Keywords: Influenza; Influenza A; Flu; Flu A
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; MEDI8852

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be assigned to Part 1 of the study (Cohort 1) in an unblinded manner.
  Part 2 is a partial double-blind study of MEDI8852 and placebo. Because MEDI8852 and placebo are not completely indistinguishable in appearance, an unblinded investigational product manager will prepare the investigational product using a coloured sleeve to cover the infusion bag containing investigational product. An unblinded investigational product monitor will perform investigational product accountability. The unblinded personnel will not reveal the treatment allocation to the sponsor or site staff. Neither the subject/legal representative nor any of the investigator or sponsor staff who are involved in the treatment or clinical evaluation of the subjects will be aware of the treatment received. In the event that the treatment allocation for a subject becomes known to the investigator or other study staff involved in the management of study subjects, the sponsor must be notified immediately.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MEDI8852 (dose 1) - part 1 (Experimental): Participants will receive a single intravenous infusion (IV) of MEDI8852 (dose 1)
  Interventions: Biological: MEDI8852
- Placebo - part 2 (Sham Comparator): Participants will received a single IV infusion of placebo ( matched to MEDI8852) on day 2
  Interventions: Drug: Placebo
- Oseltamivir (OS) 75 mg - part 2 (Active Comparator): Participants will receive 75 mg orally twice a day for 5 days starting at day 2
  Interventions: Drug: Oseltamivir
- MEDI8852 (dose 2) - part 2 (Experimental): Participants will receive a single IV dose of MEDI8852 on day 2 (dose 2)
  Interventions: Biological: MEDI8852
- MEDI8852 (dose 1) - part 2 (Experimental): Participants will receive a single IV infusion of MEDI8852 on day 2 (dose 1)
  Interventions: Biological: MEDI8852
- MEDI8852 (dose 2) +OS 75 mg part 2 (Experimental): Participants will receive a single IV infusion of MEDI8852 (dose 2) on day 2 and 75mg of Oseltamivir twice a day for 5 days starting at day 2
  Interventions: Drug: Oseltamivir; Biological: MEDI8852

INTERVENTIONS:
Drug: Oseltamivir — 75 mg capsules orally twice a day from Day 2 to Day 7
  Arms: MEDI8852 (dose 2) +OS 75 mg part 2; Oseltamivir (OS) 75 mg - part 2
Biological: MEDI8852 — MEDI8852 is a human IgG1 kappa monoclonal antibody administered as a single IV infusion at either dose 1 or dose 2 on Day 2.
  Arms: MEDI8852 (dose 1) - part 1; MEDI8852 (dose 1) - part 2; MEDI8852 (dose 2) +OS 75 mg part 2; MEDI8852 (dose 2) - part 2
Drug: Placebo — Placebo is salt-water solution containing no active ingredients and administered as a single IV infusion on Day 2.
  Arms: Placebo - part 2

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of MEDI8852 for the treatment of influenza caused by a wild type A/H1N1 challenge strain in healthy, influenza serosusceptible adults.

DETAILED DESCRIPTION:
The study will be conducted in two parts:

Part 1:

In Part 1, eight healthy subjects, 18 to 65 years of age, will be enrolled at one study center in the United States of America (USA) and will receive a single intravenous (IV) dose of MEDI8852 (Cohort 1, dose 1) on Day 1. The subjects will be admitted to a Phase 1 unit (Day -1), for dosing (Day 1) and for follow-up (through discharge from the Phase 1 unit on Day 2). Subjects will then be followed through Day 60 for treatment emergent adverse events (TEAEs), treatment emergent serious adverse events (TESAEs), treatment emergent adverse events of special interest (TEAESI), concomitant medications, nasal and blood PK, and ADA. Initiation of Part 2 of the study will be based on review of safety data from Part 1 (Days 1-8) by a study-specific Dose Evaluation Committee (DEC). For subjects in Part 1, the study is approximately 90 days in duration, consisting of a screening period of up to 30 days, a treatment period of 1 day and a follow-up period of 59 days.

Part 2:

In Part 2, approximately 60 healthy, influenza serosusceptible subjects, 18 to 65 years of age, will be enrolled at the same study center in the USA and will receive a wild-type A/H1N1 challenge strain on Day 1. Subjects will be randomized 1:1:1:1:1 into 5 cohorts (approximately 12 subjects per cohort) to receive the following on Day 2:

* Cohort 2: A single IV dose of placebo
* Cohort 3: OS, 75 mg orally BID (twice a day) for 5 days
* Cohort 4: A single IV low dose of MEDI8852 (dose 2)
* Cohort 5: A single IV high dose of MEDI8852 (dose 1)
* Cohort 6: A single IV low dose of MEDI8852 (dose 2) and oseltamivir (OS), 75 mg orally BID for 5 days

The subjects will be admitted to the Phase 1 unit (Day -1), for influenza challenge strain administration (Day 1), dosing (Day 2 [Cohorts 2, 4 and 5] and Days 2-6 [Cohorts 3 and 6]), and follow-up (through discharge from the Phase 1 unit on Day 9). Subjects will then be followed through Day 14 for solicited influenza symptoms, and through Day 60 for TEAEs, TESAEs, TEAESIs, concomitant medications, nasal and blood pharmacokinetics (PK), and antidrug antibody (ADA). For subjects in Part 2, the study is approximately 120 days in duration, consisting of a screening period of up to 60 days, a treatment period of 8 days and a follow-up period of 52 days

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 65 years at the time of screening.
* Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act [HIPAA] in the USA, European Union [EU] Data Privacy Directive in the EU) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* For subjects enrolled in Part 1 and Part 2 of the study, agree to remain restricted to an inpatient unit until released (anticipated to be 3 days and 2 nights for Part 1 and 9 days and 8 nights for Part 2).
* Able to complete the follow-up period through Day 60 as required by the protocol.
* Female subjects of childbearing potential must also have a negative urine or blood pregnancy test at screening, on Day -1 and on and Day 1 prior to randomization
* Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception for at least 2 days prior to the first dose of study drug and must agree to continue using such precautions through Day 60 of the study; cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

* History of allergic disease or reactions likely to be exacerbated by any component of the study drug, MEDI8852.
* For subjects enrolled in Part 2 of the study, history of allergic disease or reactions likely to be exacerbated by any component of OS.
* History of allergic disease or reactions to eggs or egg proteins
* Any fever ≥ 100.4°F (≥ 38.0°C) regardless of route of measurement and/or respiratory illness (eg, cough or sore throat) within 7 days prior to randomization.
* Renal impairment that would require modified dosing of OS (ie, estimated creatinine clearance of ≤ 60 mL/min).
* Any condition that, in the opinion of the investigator, might compromise subject safety or interfere with evaluation of the study drug or interpretation of subject safety or study results.
* History of Guillain-Barré syndrome.
* Hemagglutination antibody titer of >10 for the A/H1N1 challenge strain.
* Receipt of influenza antiviral therapy within the preceding 14 days.
* Concurrent participation in another interventional study.
* Previous receipt of an influenza mAb.
* Previous receipt of immunoglobulin or blood products within 6 months prior to screening.
* History of active infection with hepatitis B or C.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or serum creatinine above 1.1 times the upper limit of normal (ULN) or haemoglobin, white blood cell count, or platelet count below 0.9 times the lower limit of normal at screening.
* Known immunodeficiency due to illness, including human immunodeficiency virus infection, or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent at a dose of 20 mg daily or every other day within 6 months prior to screening.

Note: Topical corticosteroids as prescribed by a physician for an acute, uncomplicated dermatitis may be used throughout the study; over the counter medications, including topical corticosteroids for an acute, uncomplicated dermatitis, may also be used throughout the study.

* Resides in a household with an individual who has moderate to severe immunosuppression due to illness or due to drugs.

Note: Examples include individuals with symptomatic Acquired Immunodeficiency Syndrome; cancer and transplant patients who are taking immunosuppressive drugs; and those with inherited diseases that affect the immune system (e.g., congenital agammaglobulinemia, congenital IgA deficiency)

* History of chronic lung disease (eg, asthma/reactive airway disease and chronic obstructive pulmonary disease).

Note: Childhood asthma that has not required treatment in adulthood is not necessarily exclusionary

* Pregnant or nursing mother.
* History of significant cardiac disease (eg, myocarditis, pericarditis, congestive heart failure, clinically significant arrhythmias).
* History of alcohol or drug abuse within the past 2 years that, according to the investigator, might affect assessments of safety or ability of subject to comply with all study requirements.
* Any planned surgical procedure before completion of Day 60.
* Employees of the sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-03 (Estimated); Primary Completion 2020-10-09 (Estimated); Study Completion 2020-10-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of solicited influenza symptoms, treatment emergent adverse events (TEAEs), treatment emergent serious adverse events (TESAEs) and treatment emergent adverse events of special interest (TEASIs) - part 1 | Through Day 60
  To evaluate the safety and tolerability of MEDI8852 in healthy adults and influenza serosusceptible adults challenged with a wild-type A/H1N1 influenza strain
Quantification of influenza viral shedding (part2) by quantitative real time polymerase chain reaction (qRT-PCR) | On Days 2-9
  To evaluate the impact of MEDI8852, either when given alone or in combination with oseltamivir (OS), on nasal shedding of the A/H1N1 challenge strain in healthy, influenza serosusceptible adults, by qRT-PCR

SECONDARY OUTCOMES:
Time to resolution of influenza symptoms | Through Day 14
  To evaluate the effect of MEDI8852, either given alone or in combination with OS, on the time to resolution of influenza symptoms in healthy, influenza serosusceptible adults challenged with a wild-type A/H1N1 influenza strain
Relationship between the influenza viral shedding measured by quantitative real time polymerase chain reaction (qRT-PCR) and administered dose described by a dose-response model | Through Day 9
  To evaluate the effect of MEDI8852 administered at different dose levels on nasal shedding of the A/H1N1 challenge strain in healthy, influenza serosusceptible adults. An MCP-Mod statistical model will be fitted to the collected data to quantify the treatment effect in terms of viral shedding
Incidence of solicited influenza symptoms, TEAEs, TESAEs, and TEAESIs | Through Day 14 ( solicited influenza symptoms) and Through Day 60 (TEAEs, TESAEs, and TEAESIs)
  To evaluate the safety and tolerability of MEDI8852 in healthy, influenza serosusceptible adults challenged with a wild-type A/H1N1 influenza strain
MEDI8852 serum concentration | Through Day 60
  To evaluate the serum concentration of MEDI8852 in healthy adults and healthy, influenza serosusceptible adults challenged with a wild-type A/H1N1 influenza strain
The incidence of Antidrug Antibody (ADA) to MEDI8852 as summarized by the number and percentage of subjects who are ADA positive by treatment group and time point | Through Day 60
  To evaluate development of ADA to MEDI8852 from baseline through the end of the study in healthy adults, and healthy, influenza serosusceptible adults challenged with a wild-type A/H1N1 influenza strain
MEDI8852 nasal concentration | Through day 60
  To evaluate the nasal concentration of MEDI8852 in healthy adults and healthy, influenza serosusceptible adults challenged with a wild-type A/H1N1 influenza strain